CLINICAL TRIAL: NCT02755311
Title: Liver Resection Versus Transarterial Chemoembolization for the Treatment of Intermediate-stage Hepatocellular Carcinoma: a Prospective Non-randomized Trial
Brief Title: Liver Resection Versus Transarterial Chemoembolization for the Treatment of Intermediate-stage Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 006
Record Dates: First submitted 2016-04-03; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Carboplatin; Ethiodized Oil; Epirubicin; pirarubicin; hydroxycamptothecinum; Fluorouracil

ARMS (2):
- liver resection (Experimental): Resection was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant and the possibility of a negative resection margin. The investigators performed anatomical resection aiming at a resection margin of at least 1 cm. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 minutes and 5 minutes, respectively. Hemostasis of the raw liver surface was done with suturing and application of fibrin glue.
  Interventions: Procedure: liver resection
- transarterial chemoembolization (Active Comparator): A microcatheter was inserted into the feeding arteries as selectively as possible through the lobar, segmental, or subsegmental arteries, dependent on the tumor distribution and hepatic functional reserve. Hepatic artery infusion chemotherapy was performed using 300 mg carboplatin. Subsequently, chemolipiodolization was performed mixed with 5 ml of lipiodol. According to the number and size of the lesions, and liver and kidney function of the patient, the chemotherapeutic agents, including epirubicin (50-100 mg), pirarubicin (30-50 mg), hydroxycamptothecin (10-30 mg) and fluorouracil (500-1000 mg), were determined by the multidisciplinary team. If residual flow remained after infusion of these agents, additional lipiodol was injected. Embolization was performed with absorbable gelatin sponge particles 350-560 μm in diameter.
  Interventions: Procedure: transarterial chemoembolization; Drug: carboplatin; Drug: lipiodol; Drug: epirubicin , pirarubicin , hydroxycamptothecin and fluorouracil; Other: absorbable gelatin sponge particles

INTERVENTIONS:
Procedure: liver resection — Intraoperative ultrasound was routinely used during surgery. Anatomic resection was carried out in the form of segmentectomy or/and subsegmentectomy.In segmentectomy, the hepatic parenchyma was transacted at the intersegmental plane as described by Couinaud. If the hepatic parenchymal transaction plane needed to go beyond the intersegmental plane to achieve the desired extent of resection margin, the small portal branches supplying the liver parenchyma up to the intended transaction plane were punctured under US guidance and injected with methylthioninium chloride, and then liver subsegmentectomy was performed either alone or in combination with segmentectomy along the plane of demarcation as delineated by the injected methylthioninium chloride. Nonanatomic resection with a negative resection margin was performed when anatomical resection may cause inadequate liver remnant. Pringle's maneuver was used if necessary with a clamp/unclamp time of 10 min/5 min.
  Other Names: Hepatectomy
  Arms: liver resection
Procedure: transarterial chemoembolization — A microcatheter was inserted into the feeding arteries as selectively as possible through the lobar, segmental, or subsegmental arteries, dependent on the tumor distribution and hepatic functional reserve. Hepatic artery infusion chemotherapy was performed using 300 mg carboplatin. Subsequently, chemolipiodolization was performed mixed with 5 ml of lipiodol. According to the number and size of the lesions, and liver and kidney function of the patient, the chemotherapeutic agents, including epirubicin (50-100 mg), pirarubicin (30-50 mg), hydroxycamptothecin (10-30 mg) and fluorouracil (500-1000 mg), were determined by the multidisciplinary team. If residual flow remained after infusion of these agents, additional lipiodol was injected. Embolization was performed with absorbable gelatin sponge particles 350-560 μm in diameter.
  Other Names: chemoembolization through artery; TACE
  Arms: transarterial chemoembolization
Drug: carboplatin — Hepatic artery infusion chemotherapy was performed using 300 mg carboplatin (Bristol-Myers Squibb, New York, NY).
  Other Names: a drug derived from cisplatin
  Arms: transarterial chemoembolization
Drug: lipiodol — Chemolipiodolization was performed mixed with 5 ml of lipiodol (Lipiodol Ultra-Fluide; André Guerbet Laboratories, Aulnay-sous-Bois, France).
  Arms: transarterial chemoembolization
Drug: epirubicin , pirarubicin , hydroxycamptothecin and fluorouracil — The chemotherapeutic agents, including epirubicin (50-100 mg), pirarubicin (30-50 mg), hydroxycamptothecin (10-30 mg) and fluorouracil (500-1000 mg), were determined by the multidisciplinary team.
  Other Names: epirubicin，pirarubicin，hydroxycamptothecin or fluorouracil
  Arms: transarterial chemoembolization
Other: absorbable gelatin sponge particles — Embolization was performed with absorbable gelatin sponge particles (Gelfoam; Hangzhou Bi-Trumed Biotech Co., Ltd., Hangzhou, Zhejiang, China) 350-560 μm in diameter.
  Arms: transarterial chemoembolization

SUMMARY:
The role of transarterial chemoembolization (TACE) as the standard therapy for intermediate-stage hepatocellular carcinoma (HCC) is being challenged by increasing studies which showed that liver resection (LR) is a safe and feasible procedure with better survival outcomes than TACE does.

In light of this, the investigators have constructed a Markov model to simulate comparing LR and TACE in the treatment of intermediate-stage HCC. The results suggested that LR may provide survival benefit over TACE for the treatment of intermediate-stage HCC in cirrhotic patients. However, validating the simulated result by a study with higher quality (e.g. prospective clinical trial) would be of great value in providing a more convincing finding. Therefore, based on the established Markov model, the investigators aimed to prospectively compare the treatment efficacy and safety of LR with TACE for consecutive patients with intermediate-stage HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the 5th most common cancer worldwide and the third most frequent cause of death of cancer. However, the management strategies for intermediate-stage HCC remain controversial without global consensus. On one hand, Barcelona Clinic Liver Cancer (BCLC) staging system recommends liver resection (LR) for very early and early-stage HCC, and transarterial chemoembolization (TACE) for intermediate-stage HCC. On the other hand, observational studies in both Eastern and Western countries have emerged to suggest that LR was safe and achieved better survival than TACE for patients with intermediate-stage HCC, but only very few studies have been conducted to directly compare LR with TACE for these patients.

In light of this, the investigators have conducted a multistate Markov model simulating a randomized clinical trial comparing LR with TACE over a follow-up period of 15 years. The results suggested that LR may provide survival benefit over TACE for the treatment of intermediate-stage HCC in cirrhotic patients. However, validating the simulated result by a study with higher quality (e.g. prospective clinical trial) would be of great value in providing a more convincing finding.Therefore, based on the established Markov model,the investigators aimed to prospectively compare the treatment efficacy and safety of LR with TACE for consecutive patients with intermediate-stage HCC.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* 2 to 3 lesions with at least one >3 cm in diameter; or more than 3 lesions of any diameter
* Child-Pugh A/B liver function
* no previous treatment
* an Eastern Cooperative Oncology Group performance status of 0

Exclusion Criteria:

* radiologic or pathological evidence of vascular invasion or extrahepatic metastases
* severe coagulopathy (prothrombin activity <40% or a platelet count of<40,000/mm3)
* evidence of hepatic decompensation including refractory ascites, esophageal or gastric variceal bleeding, or hepatic encephalopathy
* obstructive jaundice
* an American Society of Anesthesiologists score of 3 or more
* present or past history of any other concurrent malignancies
* complicated with other severe diseases such as chronic kidney disease, cardiovascular disease, auto-immunological disease, etc
* contraindications to carboplatin, epirubicin, mitomycin, or lipiodol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  1-year overall survival

SECONDARY OUTCOMES:
Mortality | 1 month
  1-month mortality

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China